CLINICAL TRIAL: NCT07304739
Title: A Single-Arm Clinical Study of Furmonertinib (160mg) Combined With Intrathecal Chemotherapy (ITC) and Stereotactic Radiotherapy (SRT) as First-Line Treatment in EGFR Classic Mutation-Positive NSCLC Patients With Brain Parenchymal and Leptomeningeal Metastases
Brief Title: Furmonertinib Combined With Intrathecal Chemotherapy and Stereotactic Radiotherapy (SRT) for EGFR-Mutated NSCLC Patients With Brain Parenchymal and Leptomeningeal Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20250589
Record Dates: First submitted 2025-09-23; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; EGFR mutation; Brain parenchymal and meningeal metastases; Furmonertinib; Intrathecal chemotherapy; Stereotactic radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis | interventions — aflutinib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib combined with intrathecal chemotherapy and stereotactic radiotherapy group (Experimental)
  Interventions: Drug: Furmonertinib; Drug: Intrathecal chemotherapy; Radiation: Stereotactic radiotherapy

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib: 160mg, once daily, orally.
Drug: Intrathecal chemotherapy — Intrathecal chemotherapy with 40mg of pemetrexed and 2mg of dexamethasone, every 3 weeks as one cycle.
Radiation: Stereotactic radiotherapy — After two cycles of intrathecal chemotherapy, there was no progression upon re-examination. The stereotactic radiotherapy (SRT) for brain metastases with 7-19Gy/1-5Fx.

SUMMARY:
A Single-Arm Clinical Study of Furmonertinib (160mg) Combined with Intrathecal Chemotherapy (ITC) and Stereotactic Radiotherapy (SRT) as First-Line Treatment in EGFR Classic Mutation-Positive NSCLC Patients with Brain Parenchymal and Leptomeningeal Metastases

DETAILED DESCRIPTION:
The incidence of central nervous system (CNS) metastases in NSCLC representing a primary cause of mortality. In recent years, the widespread use of epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs) has significantly prolonged survival in lung adenocarcinoma patients, consequently leading to increased incidence of brain metastases (BM) and leptomeningeal metastases (LM). Both BM and LM are associated with poor prognosis. Therefore, developing more effective treatment strategies for BM and LM patients has become a cutting-edge, challenging, and critically important research focus.This study aims to evaluate the efficacy and safety of Furmonertinib (160 mg) combined with intrathecal chemotherapy and stereotactic radiotherapy (SRT) in treatment-naïve EGFR-mutated NSCLC patients with concurrent parenchymal brain and leptomeningeal metastases. The objective is to explore potential survival benefits for this poor-prognosis population and provide additional clinical treatment options.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old, male or female;
* Histopathologically confirmed, unresectable, and not amenable to curative radiotherapy treatment-naïve locally advanced or metastatic lung adenocarcinoma;
* The patient was confirmed by a local laboratory to have one of the following EGFR mutations :19Del or L858R;
* The patient has not received any systemic anti-tumor treatment in the locally advanced (the researcher judged that it was not suitable for surgery or radiotherapy) or metastatic NSCLC;
* At least one measurable tumor lesion (according to RECIST1.1);
* Confirm the simultaneous presence of brain parenchymal and meningeal metastasis;
* Laboratory tests indicated that the subjects had adequate organ functions, including: 1) ANC ≥1.5×109/L; PLT ≥100×109/L; HGB ≥90g/L; 2) TBIL ≤1.5 times the upper limit of the normal value, AST and ALT ≤2.5 times the upper limit of the normal value (for those with liver metastasis, total bilirubin ≤ 3 times the upper limit of the normal value, AST and ALT≤ 5 times the upper limit of the normal value are allowed); 3) CrCL ≥50 ml/min (calculated according to the Cockcroft-Gault formula);
* The ECOG score at the time of screening was 0-2, and there was no significant deterioration of the disease within 2 weeks before the screening;
* The expected survival period is greater than 12 weeks;
* Non-pregnant female patients of childbearing potential with no pregnancy plan. Female subjects of childbearing potential and male subjects must agree to use effective contraception during the study period and for 6 months after discontinuation of the study drug;
* Understand and voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* Histological or cytological examination suggests NSCLC dominated by squamous cells, or indicates the presence of small cell lung cancer, neuroendocrine carcinoma, etc.；
* Patients with other driver genes: ALK, ROS1, RET, BRAF, NTRK, MET, KRAS, etc.. But TP53, RB1, BRAC are not included；
* Anticipated requirement for other antitumor therapies beyond this clinical trial during the study period;
* Having received any of the following treatments: a) Major surgery within 4 weeks prior to the first dose or during the trial period, excluding procedures such as vascular access establishment, mediastinoscopy, or thoracoscopy for biopsy; b) Use of strong CYP3A4 inhibitors within 7 days or strong CYP3A4 inducers within 21 days prior to the first dose; Use of Chinese herbal medicines or preparations with anti-tumor indications or those adjunctive to cancer therapy within 2 weeks prior to the first dose or expected during the trial period; c) Participation in an investigational drug or device clinical trial within 4 weeks or at least 5 half-lives (whichever is longer) prior to the first dose; d) Treatment with other antitumor drugs within 14 days prior to the first dose;
* Patients with symptomatic and unstable pleural or peritoneal effusion; those who have achieved clinical stability for at least 14 days after drainage of pleural effusion or ascites may be enrolled;
* Toxicities from prior antitumor therapy have not recovered to ≤ CTCAE grade 1(with the exception of alopecia and residual neurotoxicity from previous platinum-based therapy)；
* History of other malignancies or currently concurrent other malignancies (except for malignancies that have undergone radical resection with no recurrence within 5 years, such as cervical carcinoma in situ, basal cell carcinoma of the skin, and papillary thyroid carcinoma);
* History of interstitial lung disease (ILD), drug-induced ILD, or radiation pneumonitis requiring steroid treatment; or current clinical manifestations suggestive of ILD;
* Severe or uncontrolled systemic diseases requiring treatment including hypertension, diabetes, chronic heart failure (NYHA class III-IV), unstable angina, myocardial infarction within the past year, active hemorrhagic conditions, severe gastrointestinal disorders, active infectious diseases, etc.;
* Resting QT interval (QTc) > 470 msec as measured by clinical ECG screening; Clinically significant prolonged QT interval or other arrhythmias or clinical conditions that may increase the risk of QT prolongation;
* Known history of psychiatric disorders or drug abuse, with current active symptoms or ongoing drug use;
* Known or suspected hypersensitivity to furmonertinib or any excipients of its formulation;
* Female subjects who are pregnant or breastfeeding, or female partners of male subjects who plan to become pregnant during the study period;
* The subject demonstrated poor compliance;
* Any other condition deemed by the investigator to make the subject unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
iPFS | From enrollment to the occurrence of intracranial disease progression (excluding non-intracranial progression) or death，assessed up to 2 year
  iPFS is defined as the time from the start of treatment to the occurrence of intracranial disease progression (excluding non-intracranial progression) or death

SECONDARY OUTCOMES:
PFS | from the start of treatment to the occurrence of tumor progression or all-cause death, assessed up to 2 year
  defined as the time from the start of treatment to the occurrence of objective tumor progression or all-cause death
OS | from the start of treatment to death, 2 years
LM remission rate | Until the end of the study, 1year
iORR | From enrollment to the end of treatment at 1 year
  The proportion of patients achieving a pre-specified reduction in intracranial lesion volume sustained for the minimum required duration (at least 4 weeks).
iDCR | From enrollment to the end of treatment at 1year
  The proportion of subjects with intracranial lesions achieving disease control (including complete response [CR], partial response [PR], or stable disease [SD]) from the initiation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maobin Meng, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (3):
- China (3):
  - CANGZHOU People's Hospital, Cangzhou, Hebei
  - Tianjin medical university cancer hospital and institute, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No